CLINICAL TRIAL: NCT04444245
Title: Re-establishment of Ovarian Hormonal Function, Delay of Menopause, or Reversal of Early Menopause With High Density (HD PRP), tSVF + PRP, or Cell Enriched tSVF + PRP by Ultrasound Guided Ovarian Injection
Brief Title: Ovarian Rejuvenation Using Platelet Rich Plasma (PRP) & Autologous Tissue Stromal Vascular Fraction (tSVF) and Cell Enriched tSVF
Acronym: OVAR-REJUV
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Black Tie Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVARIAN REJUV
Record Dates: First submitted 2020-06-02; First posted 2020-06-23 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Ovarian Failure; Perimenopausal Disorder; Hormone Disturbance
MeSH Terms: conditions — Endocrine System Diseases | interventions — Saline Solution; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ARM 1 Platelet Rich Plasma (Experimental): Blood draw, processing of PRP, white blood cell poor, high platelet multiple >/= 4, e.g. (Emcyte II Pure PRP) Endovaginal ultrasound guided intra-ovarian placement into ovarian parenchyma, preferably both if accessible.
  Interventions: Procedure: lipoaspiration harvest tSVF; Procedure: Platelet Rich Plasma; Procedure: Endovaginal Ultrasound
- ARM 2 emulsified tSVF and PRP (Experimental): Blood draw, processing of PRP, white blood cell poor, high platelet multiple >/= 4, e.g. Emcyte PRP Lipoaspiration utilizing closed microcannula harvesting of small volume (Tulip tumescent fluid infiltrator and Tulip Harvester). Decanting of free lipid. Emulsification of adipose tissue into tSVF (Tulip Nanofat device). Blending of Nanofat with PRP at a 3:1 ratio.
  Endovaginal ultrasound guided intra-ovarian placement into ovary, preferably both if accessible.
  Interventions: Procedure: lipoaspiration harvest tSVF; Procedure: Platelet Rich Plasma; Procedure: Endovaginal Ultrasound; Drug: Normal Saline (NS) .9% 10 mL Injection; Device: emulsification tSVF
- ARM 3 emulsified tSVF and PRP, enriched with cSVF (Experimental): Blood draw, processing of PRP, white blood cell poor, high platelet multiple >/= 4, e.g. Emcyte PRP tSVF preparation: Lipoaspiration utilizing closed microcannula harvesting of small volume (Tulip tumescent fluid infiltrator and Tulip Harvester). Decanting of free lipid. Emulsification of adipose tissue (Tulip Nanofat device).
  cSVF preparation: lipoaspiration as above. Isolation and Concentration of cellular stromal vascular fraction (cSVF) using a Healeon Medical CentriCyte 1000 centrifuge, incubator and shaker plate with sterile Liberase enzyme (Roche Medical) per manufacturer protocol. Quantification of viable nucleated cell count with flow cytometry. Addition of pellet of viable nucleated cells to tSVF.
  Blending of tSVF/cSVF emulsion with PRP at a 3:1 ratio. Endovaginal ultrasound guided intra-ovarian placement into ovary, preferably both if accessible.
  Intervention:
  Interventions: Procedure: lipoaspiration harvest tSVF; Procedure: Platelet Rich Plasma; Procedure: Endovaginal Ultrasound; Device: Cellular Isolation cSVF; Drug: Normal Saline (NS) .9% 10 mL Injection; Device: emulsification tSVF
- ARM 4 Intra-ovarian guided placement (Experimental): Specifically designed 23 gauge modified oocyte harvester needle for ultrasound guided placement
  Interventions: Procedure: Endovaginal Ultrasound

INTERVENTIONS:
Procedure: lipoaspiration harvest tSVF — Use of disposable, sterile microcannula lipoharvest to acquire tSVF
  Arms: ARM 1 Platelet Rich Plasma; ARM 2 emulsified tSVF and PRP; ARM 3 emulsified tSVF and PRP, enriched with cSVF
Procedure: Platelet Rich Plasma — Standard venipuncture, concentration of PRP in FDA approved device (Emcyte II)
  Arms: ARM 1 Platelet Rich Plasma; ARM 2 emulsified tSVF and PRP; ARM 3 emulsified tSVF and PRP, enriched with cSVF
Procedure: Endovaginal Ultrasound — Endovaginal Ultrasound guidance to intra-ovarian placement, bilaterally
Device: Cellular Isolation cSVF — Digestion of tSVF with Liberase, isolation & concentration of cSVF in Centricyte 1000
  Arms: ARM 3 emulsified tSVF and PRP, enriched with cSVF
Drug: Normal Saline (NS) .9% 10 mL Injection — 10 cc Sterile Normal Saline for Injection
  Arms: ARM 2 emulsified tSVF and PRP; ARM 3 emulsified tSVF and PRP, enriched with cSVF
Device: emulsification tSVF — Harvested tSVF emulsification with sterile, disposable Nanofat screen device
  Arms: ARM 2 emulsified tSVF and PRP; ARM 3 emulsified tSVF and PRP, enriched with cSVF

SUMMARY:
Trial of imaging guided intra-ovarian injection to improve ovarian function in clinical settings of Premature Ovarian Failure, Perimenopausal and /or early postmenopausal symptomatology and related hormonal deficiencies. The study will compare the effectiveness of autologous Platelet Rich Plasma alone versus Stromal Vascular Fraction (tSVF and/or cellular stromal vascular fraction (cSVF) in combination with Platelet Rich Plasma as regards efficacy and duration of ovarian reactivation in women with acquired Premature Ovarian Failure, Menopausal, and Perimenopausal women.

DETAILED DESCRIPTION:
Intra-ovarian placement of platelet rich plasma (PRP) has already been demonstrated in several series to return peri-menopausal and early post-menopausal hormone levels towards pre-menopausal levels and pre-menopausal cyclic behavior, even resulting in pregnancies and deliveries of healthy infants. The intent of this trial is to evaluate the utility of PRP to improve hormonal status and clinical symptomatology in peri-menopausal and early post-menopausal women, and in women with non-Turner's premature ovarian failure, by documenting the improvements in biochemical/hormonal parameters, bone density, and physical and mental health related quality of life, as well as comparing the duration and effectiveness of this PRP procedure with the intra-ovarian placement of biocellular physiologically active cellular and cytokine elements contained within the adipose tissue-derived Stromal Vascular Fraction (tSVF).

It should be noted that rate of loss of bone density in women is maximal in the 12 months prior and 24 months following menopause. The absolute and relative percentage amounts of body fat and muscle change in adverse ways - with increasing fat and falling muscle bulk, with the most dramatic changes also occurring in the menopausal transition period. This study therefore provides the potential to document measurable cessation of bone density loss or reduction in rate of bone density loss compared to well established known patterns and historical controls as a result of the proposed relatively innocuous interventions. The same technology to be used for bone density evaluation, single photon absorptiometry, will also be used to quantify fat versus muscle body composition at baseline and 18 months.

SVF can be further characterized as either cellular SVF or tissue SVF (cSVF or tSVF). Tissue SVF (tSVF) is obtained by a small volume manual closed syringe microcannula aspiration of subcutaneous fatty tissue (approximately 10+ teaspoons), followed by closed system decanting to remove the infranatant fluids followed by emulsification of the remnant to the required degree of homogeneity and reduced particulate size to permit injection through a conventional gauge needle bores. Tissue SVF is characterized by retention of a proportion of the non-cellular matrix of collagenous and fine vascular remnants, which together form a matrix that retains and provides structure to the biocellular elements that are embedded within. Cellular SVF (cSVF) begins with the same mini-aspiration, but is characterized by closed system centrifugation, followed enzymatic digestion to isolate./concentrate the cellular SVF (cSVF). Following enzyme neutralization and rinsing, the resultant concentrate of viable stem/stromal nucleated cells, are prepared for guided placement into the ovarian parenchymal tissue. A sample of each injectate is tested and quantified using standard laser flow cytometry, including viability and numbers of cells within each sample.

The study includes use of PRP (Emcyte II Pure PRP, Florida, USA) PRP per manufacturer's instructions) alone as control in first treatment limb (ARM), which will volumetrically be the same as the other injectates, for guided placement documented within the ovaries. A comparative second ARM composed of PRP will be combined with emulsified tSVF (Sterile Tulip Nanofat Disposable, San Diego, California (CA), USA) . In a third ARM, PRP plus emulsified tSVF will be combined with both concentrated cSVF. This arm is to determine effects of higher cellular concentration than achieved in second ARM using the cellular concentrates achieve using the Centricyte 1000 (Healeon Medical Inc, Newbury Park, CA, USA). The primary outcomes for each of these optional procedures will be compared, and evaluated as to safety, clinical efficacy in enhancing return of ovarian function to determine the preferred methodology to achieve maximal outcomes.

Baseline and monitored patient characteristics are as follows:

* Baseline status of all patients will determined utilizing relevant biochemical indices, including serum levels of Follicle Stimulating Hormone (FSH), Anti-Mullerian Hormone (AMH), Luteinizing Hormone (LH), Estradiol (E2), and Progesterone (PRG). These will be repeated at 30 and 90 days, and then every 3 months for an additional 15 months, total follow up 18 months. Comprehensive Blood Panel (SMA 12), Complete blood count (CBC), lipid profiles and clotting indices will be obtained at baseline and repeated (without clotting indices) at 12 months.
* As bone density begins to decline at a significant rate in the peri-menopausal period, a bone density determination with single photon absorptiometry will be obtained at baseline, and again at 12 and/or 18 months. Body composition fat/muscle proportions will be evaluated with the same technology at the same sitting.
* Physical and mental health related quality of life will be evaluated with the quality of life surveys at baseline, 6 and 12 months.
* Ovarian volume will be assessed at baseline by endovaginal sonography, along with the size and number of follicles present, and then every 6 months.
* Journal recording of menstrual cycles - frequency/interval, days, and duration.

In ARM 1, PRP alone will be placed within the ovaries. In ARM 2, PRP will be combined with tSVF. In ARM 3, tSVF will be combined with both cSVF and PRP. Matched volumes of injectate will be used in each ARM to avoid question of potential interference to ovarian parenchyma impacting the outcome due to volume variable effects. The primary outcomes for each of these arms will be compared, informing us of a preferred methodology for further evaluation, and ultimately, clinical practice.

Autologous Platelet Rich Plasma is an established treatment modality which utilizes FDA approved methodologies and kits, and has developed into a mature treatment modality for a variety of orthopedic and soft tissue pathologies. As noted, its safety and utility in ovarian rejuvenation and reversal of infertility has already been established in peer reviewed, case series.

Safety of use of certain allogeneic human mesenchymal stem cells (hMSC) has been proposed and limitedly tested for efficacy in some prior studies. The products tested have variable protocols in isolating and documenting content and cellular viabilities.

Autologous stem-stromal cells (contained within cSVF) have been reported safe and effective in many applications/studies and in clinical trials currently underway in other body systems and pathologies. These cells are easily obtained and isolated/concentrated in a closed system from patient's adipose derived stromal vascular fraction (tSVF). This is important as such tissues are the patient's own, genetically unique cells and, in theory, potentially safer than the allogeneic human mesenchymal stem cells (hMSCs) which are potentially genetically foreign and bear the risk of contamination in processing and delivery.

A combined approach may allow the implementation of a suitably larger number of cells, growth factors, exosomes/microvesicles without the need for culture expansion.

Contents of the cSVF contains a heterogeneous population of undesignated (stem-like) and supportive cells (stromal). This combination of adult, autologous cells, along with stromal cells are felt to offer important therapeutic and regenerative qualities based cellular differentiation features and the paracrine (secretory communication signals and responses to niche) in varying degrees. It is believed that such signaling may constitute the body's own mechanism for homeostasis and regeneration. Interaction of these complex biochemical signals, are proposed to further recruit or activate reparative processes with interaction with the native host cells and tissues. Furthermore, this reparative process may become important specific host activities and needs in the location into which the therapeutic combination is placed. The precise mechanisms underlying these reparative processes are under intensive investigations.

In all cases, the platelet and biocellular materials for intra-ovarian injection will be placed under conventional imaging guidance utilizing endovaginal sonography. Specially designed modified needles will be utilized to accurate deliver the biological products to the targeted intra-ovarian parenchymal tissues. The methodology required is very similar overall to oocyte retrieval in infertility treatments, which are performed worldwide, with minimal risk of adverse effects millions of times every year.

The procedures are known to result in minimal discomfort,with patient preparation varying from none to mild supportive anxiolysis. Post procedure pain, if any, can be effectively managed with acetaminophen. Patients are observed post procedure for 60-120 minutes, and then discharged with suitable post-procedure written instructions to periodically return for clinical and laboratory follow up per protocol outlined in the outcomes analysis. The goal of this study seeks to compare the duration of hormonal, clinical, and quality of life improvement among the 3 arms of the study.

For the minority of study participants in whom ovaries are not readily accessible by endovaginal ultrasound, a subset of patients may require use of laparoscopic guidance. In all such cases, the interventions will take place in hospital settings, with the Investigator preparing the injectate and gynecologic or other suitable specialist surgeons performing the laparoscopic procedure utilizing standard procedures as the guidance.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatology or hormonal derangement for at least 6 months
* Stopped Hormonal Replacement Therapy (HRT) for at least 3 months prior to intervention
* Stopped Botanotherapy / Danazol for 3 months
* Willing to comply with study requirements, including avoiding HRT, Botanotherapy, Danazol for at least 12 months post intervention.
* Women over the age of 35
* Presence of at least one ovary
* Agree to report any pregnancy to the research staff immediately.
* Willing and able to comply with study requirements.

Exclusion Criteria:

* Current or previous Immune Globulin A (IgA) deficiency
* Current or previous premature ovarian failure due to a genetic origin, such as Turner's Syndrome or chromosomal abnormality
* Current or previous injuries or adhesions to the pelvis or ovaries
* Current and ongoing pregnancy
* Current and ongoing anticoagulant use
* Known bleeding diathesis
* Current and ongoing major Mental health disorder that precludes participation in the study
* Current and ongoing active substance abuse or dependence
* Prior or current ovarian malignancy, or known genetic mutation
* Current and ongoing chronic pelvic pain other than dyspareunia or vulval/vaginal integument disorders
* History of endometriosis
* Current diagnosis of cancer or active cancer within last 24 months
* Ovarian inaccessibility determined by endovaginal sonography
* Current or previous premature ovarian failure
* Active, untreated Endocrinologic disorders (uncompensated thyroid dysfunction, insulin dependant diabetes (type 1, type2)
* Body Mass Index (BMI) >30 kg/m2
* Systemic autoimmune disorder
* Know Polycystic Ovarian Syndrome
* Unwilling to terminate ovarian pharmaceuticals or exogenous hormone treatments 3 months prior to entering study, and to avoid exogenous hormones for duration of study

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Ovaries must be present.
Enrollment: 100 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Patient Safety For Procedure | 30 days
  Reporting of all Adverse Events, Severe Adverse Events

SECONDARY OUTCOMES:
Menstrual Resumption | baseline through 18 months
  Journal documentation by subjects of menstrual frequency, duration
Hormonal Response | Baseline, 3 months, 6 months, 12 months, 18 months
  Concentrations of Follicular Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol, Anti-Mullerian Hormone. Percentage of patients with significant reductions in FSH and LH, increases in Estradiol and Anti-Mullerian Hormone will be tabulated. Changes in these directions will indicate improved hormonal status that has been shown to correlate with improved health status across a wide range of measures.
Ovarian Morphology | Baseline, 6 month, 12 month, 18 month
  Endovaginal Sonography for Ovarian Volume
Bone Density and Body Composition | Baseline, 12 and/or 18 months
  Evaluation of Bone density and Body Composition (fat /muscle proportions) by Single Photon Absorptiometry

OTHER OUTCOMES:
Health Related Quality of Life | Baseline, 6 months, 12 months
  Utian Menopausal Quality of Life (UQoL )Instrument and the SF-36v2 physical and mental health quality of life surveys. These are norm based clinically validated and widely accepted measurement tools. Improving scores would indicate increased subject satisfaction with general physical and mental health for the SF-36v2 survey, and reduced menopausal-specific symptomatology for the Utian Menopausal Quality of Life survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Fanny Island Campus Medical Building, Colchester, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He Y, Chen D, Yang L, Hou Q, Ma H, Xu X. The therapeutic potential of bone marrow mesenchymal stem cells in premature ovarian failure. Stem Cell Res Ther. 2018 Oct 4;9(1):263. doi: 10.1186/s13287-018-1008-9. PMID 30286808
- [Background] Sills ES, Rickers NS, Li X, Palermo GD. First data on in vitro fertilization and blastocyst formation after intraovarian injection of calcium gluconate-activated autologous platelet rich plasma. Gynecol Endocrinol. 2018 Sep;34(9):756-760. doi: 10.1080/09513590.2018.1445219. Epub 2018 Feb 28. PMID 29486615
- [Background] Bertone-Johnson ER, Manson JE, Purdue-Smithe AC, Steiner AZ, Eliassen AH, Hankinson SE, Rosner BA, Whitcomb BW. Anti-Mullerian hormone levels and incidence of early natural menopause in a prospective study. Hum Reprod. 2018 Jun 1;33(6):1175-1182. doi: 10.1093/humrep/dey077. PMID 29659835
- [Background] Ji MX, Yu Q. Primary osteoporosis in postmenopausal women. Chronic Dis Transl Med. 2015 Mar 21;1(1):9-13. doi: 10.1016/j.cdtm.2015.02.006. eCollection 2015 Mar. No abstract available. PMID 29062981
- [Background] Li J, Yu Q, Huang H, Deng W, Cao X, Adu-Frimpong M, Yu J, Xu X. Human chorionic plate-derived mesenchymal stem cells transplantation restores ovarian function in a chemotherapy-induced mouse model of premature ovarian failure. Stem Cell Res Ther. 2018 Apr 3;9(1):81. doi: 10.1186/s13287-018-0819-z. PMID 29615109
- [Background] Liu M, Qiu Y, Xue Z, Wu R, Li J, Niu X, Yuan J, Wang Y, Wu Q. Small extracellular vesicles derived from embryonic stem cells restore ovarian function of premature ovarian failure through PI3K/AKT signaling pathway. Stem Cell Res Ther. 2020 Jan 3;11(1):3. doi: 10.1186/s13287-019-1508-2. PMID 31900201
- [Background] Vermeulen M, Giudice MG, Del Vento F, Wyns C. Role of stem cells in fertility preservation: current insights. Stem Cells Cloning. 2019 Aug 5;12:27-48. doi: 10.2147/SCCAA.S178490. eCollection 2019. PMID 31496751
- [Background] Zhang X, Niu J, Che T, Zhu Y, Zhang H, Qu J. Fertility preservation in BRCA mutation carriers-efficacy and safety issues: a review. Reprod Biol Endocrinol. 2020 Feb 18;18(1):11. doi: 10.1186/s12958-019-0561-0. PMID 32070378
- [Background] Ling L, Feng X, Wei T, Wang Y, Wang Y, Wang Z, Tang D, Luo Y, Xiong Z. Human amnion-derived mesenchymal stem cell (hAD-MSC) transplantation improves ovarian function in rats with premature ovarian insufficiency (POI) at least partly through a paracrine mechanism. Stem Cell Res Ther. 2019 Jan 25;10(1):46. doi: 10.1186/s13287-019-1136-x. PMID 30683144
- [Background] Su J, Ding L, Cheng J, Yang J, Li X, Yan G, Sun H, Dai J, Hu Y. Transplantation of adipose-derived stem cells combined with collagen scaffolds restores ovarian function in a rat model of premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):1075-86. doi: 10.1093/humrep/dew041. Epub 2016 Mar 9. PMID 26965432
- [Background] Zhao YX, Chen SR, Su PP, Huang FH, Shi YC, Shi QY, Lin S. Using Mesenchymal Stem Cells to Treat Female Infertility: An Update on Female Reproductive Diseases. Stem Cells Int. 2019 Dec 6;2019:9071720. doi: 10.1155/2019/9071720. eCollection 2019. PMID 31885630
- [Background] Liu R, Zhang X, Fan Z, Wang Y, Yao G, Wan X, Liu Z, Yang B, Yu L. Human amniotic mesenchymal stem cells improve the follicular microenvironment to recover ovarian function in premature ovarian failure mice. Stem Cell Res Ther. 2019 Oct 2;10(1):299. doi: 10.1186/s13287-019-1315-9. PMID 31578152
- [Background] Yoon SY. Mesenchymal stem cells for restoration of ovarian function. Clin Exp Reprod Med. 2019 Mar;46(1):1-7. doi: 10.5653/cerm.2019.46.1.1. Epub 2019 Mar 1. PMID 30827071
- [Background] Chen L, Guo S, Wei C, Li H, Wang H, Xu Y. Effect of stem cell transplantation of premature ovarian failure in animal models and patients: A meta-analysis and case report. Exp Ther Med. 2018 May;15(5):4105-4118. doi: 10.3892/etm.2018.5970. Epub 2018 Mar 20. PMID 29755593
- [Background] Tabatabaei Qomi R, Sheykhhasan M. Adipose-derived stromal cell in regenerative medicine: A review. World J Stem Cells. 2017 Aug 26;9(8):107-117. doi: 10.4252/wjsc.v9.i8.107. PMID 28928907
- [Background] Ding C, Li H, Wang Y, Wang F, Wu H, Chen R, Lv J, Wang W, Huang B. Different therapeutic effects of cells derived from human amniotic membrane on premature ovarian aging depend on distinct cellular biological characteristics. Stem Cell Res Ther. 2017 Jul 27;8(1):173. doi: 10.1186/s13287-017-0613-3. PMID 28750654
- [Background] Li F, Zhou C, Xu L, Tao S, Zhao J, Gu Q. Effect of Stem Cell Therapy on Bone Mineral Density: A Meta-Analysis of Preclinical Studies in Animal Models of Osteoporosis. PLoS One. 2016 Feb 16;11(2):e0149400. doi: 10.1371/journal.pone.0149400. eCollection 2016. PMID 26882451
- [Background] Bidet M, Bachelot A, Bissauge E, Golmard JL, Gricourt S, Dulon J, Coussieu C, Badachi Y, Touraine P. Resumption of ovarian function and pregnancies in 358 patients with premature ovarian failure. J Clin Endocrinol Metab. 2011 Dec;96(12):3864-72. doi: 10.1210/jc.2011-1038. Epub 2011 Oct 12. PMID 21994953
- [Background] Cordts EB, Christofolini DM, Dos Santos AA, Bianco B, Barbosa CP. Genetic aspects of premature ovarian failure: a literature review. Arch Gynecol Obstet. 2011 Mar;283(3):635-43. doi: 10.1007/s00404-010-1815-4. Epub 2010 Dec 29. PMID 21188402
- [Background] Miao Y, Wang P, Xie B, Yang M, Li S, Cui Z, Fan Y, Li M, Xiong B. BRCA2 deficiency is a potential driver for human primary ovarian insufficiency. Cell Death Dis. 2019 Jun 17;10(7):474. doi: 10.1038/s41419-019-1720-0. PMID 31209201
- [Background] Hernandez-Angeles C, Castelo-Branco C. Early menopause: A hazard to a woman's health. Indian J Med Res. 2016 Apr;143(4):420-7. doi: 10.4103/0971-5916.184283. PMID 27377497
- [Background] Guo Y, Sun J, Lai D. Role of microRNAs in premature ovarian insufficiency. Reprod Biol Endocrinol. 2017 May 12;15(1):38. doi: 10.1186/s12958-017-0256-3. PMID 28499456
- [Background] Chen X, Wang Q, Li X, Wang Q, Xie J, Fu X. Heat shock pretreatment of mesenchymal stem cells for inhibiting the apoptosis of ovarian granulosa cells enhanced the repair effect on chemotherapy-induced premature ovarian failure. Stem Cell Res Ther. 2018 Sep 26;9(1):240. doi: 10.1186/s13287-018-0964-4. PMID 30257708
- [Background] Vural B, Duruksu G, Vural F, Gorguc M, Karaoz E. Effects of VEGF + Mesenchymal Stem Cells and Platelet-Rich Plasma on Inbred Rat Ovarian Functions in Cyclophosphamide-Induced Premature Ovarian Insufficiency Model. Stem Cell Rev Rep. 2019 Aug;15(4):558-573. doi: 10.1007/s12015-019-09892-5. PMID 31037585
- [Background] Liu C, Yin H, Jiang H, Du X, Wang C, Liu Y, Li Y, Yang Z. Extracellular Vesicles Derived from Mesenchymal Stem Cells Recover Fertility of Premature Ovarian Insufficiency Mice and the Effects on their Offspring. Cell Transplant. 2020 Jan-Dec;29:963689720923575. doi: 10.1177/0963689720923575. PMID 32363925
- [Background] Ding C, Zou Q, Wang F, Wu H, Chen R, Lv J, Ling M, Sun J, Wang W, Li H, Huang B. Human amniotic mesenchymal stem cells improve ovarian function in natural aging through secreting hepatocyte growth factor and epidermal growth factor. Stem Cell Res Ther. 2018 Mar 9;9(1):55. doi: 10.1186/s13287-018-0781-9. PMID 29523193
- [Background] Li J, Mao Q, He J, She H, Zhang Z, Yin C. Human umbilical cord mesenchymal stem cells improve the reserve function of perimenopausal ovary via a paracrine mechanism. Stem Cell Res Ther. 2017 Mar 9;8(1):55. doi: 10.1186/s13287-017-0514-5. PMID 28279229
- [Background] Takehara Y, Yabuuchi A, Ezoe K, Kuroda T, Yamadera R, Sano C, Murata N, Aida T, Nakama K, Aono F, Aoyama N, Kato K, Kato O. The restorative effects of adipose-derived mesenchymal stem cells on damaged ovarian function. Lab Invest. 2013 Feb;93(2):181-93. doi: 10.1038/labinvest.2012.167. Epub 2012 Nov 19. PMID 23212100
- [Background] Huang B, Lu J, Ding C, Zou Q, Wang W, Li H. Exosomes derived from human adipose mesenchymal stem cells improve ovary function of premature ovarian insufficiency by targeting SMAD. Stem Cell Res Ther. 2018 Aug 9;9(1):216. doi: 10.1186/s13287-018-0953-7. PMID 30092819
- [Background] Shen J, Cao D, Sun JL. Ability of human umbilical cord mesenchymal stem cells to repair chemotherapy-induced premature ovarian failure. World J Stem Cells. 2020 Apr 26;12(4):277-287. doi: 10.4252/wjsc.v12.i4.277. PMID 32399136
- [Background] Fazeli Z, Abedindo A, Omrani MD, Ghaderian SMH. Mesenchymal Stem Cells (MSCs) Therapy for Recovery of Fertility: a Systematic Review. Stem Cell Rev Rep. 2018 Feb;14(1):1-12. doi: 10.1007/s12015-017-9765-x. PMID 28884412
- [Background] Bu S, Zhang Q, Wang Q, Lai D. Human amniotic epithelial cells inhibit growth of epithelial ovarian cancer cells via TGF-beta1-mediated cell cycle arrest. Int J Oncol. 2017 Nov;51(5):1405-1414. doi: 10.3892/ijo.2017.4123. Epub 2017 Sep 14. PMID 29048644
- [Background] Herraiz S, Pellicer N, Romeu M, Pellicer A. Treatment potential of bone marrow-derived stem cells in women with diminished ovarian reserves and premature ovarian failure. Curr Opin Obstet Gynecol. 2019 Jun;31(3):156-162. doi: 10.1097/GCO.0000000000000531. PMID 30855290
- [Background] Bhartiya D, Patel H. Ovarian stem cells-resolving controversies. J Assist Reprod Genet. 2018 Mar;35(3):393-398. doi: 10.1007/s10815-017-1080-6. Epub 2017 Nov 11. PMID 29128912
- [Background] Vanni VS, Vigano P, Papaleo E, Mangili G, Candiani M, Giorgione V. Advances in improving fertility in women through stem cell-based clinical platforms. Expert Opin Biol Ther. 2017 May;17(5):585-593. doi: 10.1080/14712598.2017.1305352. Epub 2017 Mar 28. PMID 28351161
- [Background] Farimani M, Heshmati S, Poorolajal J, Bahmanzadeh M. A report on three live births in women with poor ovarian response following intra-ovarian injection of platelet-rich plasma (PRP). Mol Biol Rep. 2019 Apr;46(2):1611-1616. doi: 10.1007/s11033-019-04609-w. Epub 2019 Feb 5. PMID 30725347
- [Background] Ruhle A, Lopez Perez R, Zou B, Grosu AL, Huber PE, Nicolay NH. The Therapeutic Potential of Mesenchymal Stromal Cells in the Treatment of Chemotherapy-Induced Tissue Damage. Stem Cell Rev Rep. 2019 Jun;15(3):356-373. doi: 10.1007/s12015-019-09886-3. PMID 30937640
- [Background] Zafardoust S, Kazemnejad S, Darzi M, Fathi-Kazerooni M, Rastegari H, Mohammadzadeh A. Improvement of Pregnancy Rate and Live Birth Rate in Poor Ovarian Responders by Intraovarian Administration of Autologous Menstrual Blood Derived- Mesenchymal Stromal Cells: Phase I/II Clinical Trial. Stem Cell Rev Rep. 2020 Aug;16(4):755-763. doi: 10.1007/s12015-020-09969-6. PMID 32198596
- [Background] Truman AM, Tilly JL, Woods DC. Ovarian regeneration: The potential for stem cell contribution in the postnatal ovary to sustained endocrine function. Mol Cell Endocrinol. 2017 Apr 15;445:74-84. doi: 10.1016/j.mce.2016.10.012. Epub 2016 Oct 12. PMID 27743990
- [Background] Sheikhansari G, Aghebati-Maleki L, Nouri M, Jadidi-Niaragh F, Yousefi M. Current approaches for the treatment of premature ovarian failure with stem cell therapy. Biomed Pharmacother. 2018 Jun;102:254-262. doi: 10.1016/j.biopha.2018.03.056. Epub 2018 Mar 22. PMID 29567538
- [Background] Soleimani R, Heytens E, Darzynkiewicz Z, Oktay K. Mechanisms of chemotherapy-induced human ovarian aging: double strand DNA breaks and microvascular compromise. Aging (Albany NY). 2011 Aug;3(8):782-93. doi: 10.18632/aging.100363. PMID 21869459
- [Background] Galvez-Martin P, Sabata R, Verges J, Zugaza JL, Ruiz A, Clares B. Mesenchymal Stem Cells as Therapeutics Agents: Quality and Environmental Regulatory Aspects. Stem Cells Int. 2016;2016:9783408. doi: 10.1155/2016/9783408. Epub 2016 Nov 24. PMID 27999600
- [Background] Wang S, Yu L, Sun M, Mu S, Wang C, Wang D, Yao Y. The therapeutic potential of umbilical cord mesenchymal stem cells in mice premature ovarian failure. Biomed Res Int. 2013;2013:690491. doi: 10.1155/2013/690491. Epub 2013 Aug 13. PMID 23998127
- [Background] Santiquet N, Vallieres L, Pothier F, Sirard MA, Robert C, Richard F. Transplanted bone marrow cells do not provide new oocytes but rescue fertility in female mice following treatment with chemotherapeutic agents. Cell Reprogram. 2012 Apr;14(2):123-9. doi: 10.1089/cell.2011.0066. PMID 22471934
- [Background] Sun M, Wang S, Li Y, Yu L, Gu F, Wang C, Yao Y. Adipose-derived stem cells improved mouse ovary function after chemotherapy-induced ovary failure. Stem Cell Res Ther. 2013 Jul 9;4(4):80. doi: 10.1186/scrt231. PMID 23838374
- [Background] Kilic S, Pinarli F, Ozogul C, Tasdemir N, Naz Sarac G, Delibasi T. Protection from cyclophosphamide-induced ovarian damage with bone marrow-derived mesenchymal stem cells during puberty. Gynecol Endocrinol. 2014 Feb;30(2):135-40. doi: 10.3109/09513590.2013.860127. Epub 2013 Dec 6. PMID 24308768
- [Background] Frese L, Dijkman PE, Hoerstrup SP. Adipose Tissue-Derived Stem Cells in Regenerative Medicine. Transfus Med Hemother. 2016 Jul;43(4):268-274. doi: 10.1159/000448180. Epub 2016 Jul 26. PMID 27721702
- [Background] Xia X, Wang T, Yin T, Yan L, Yan J, Lu C, Zhao L, Li M, Zhang Y, Jin H, Zhu X, Liu P, Li R, Qiao J. Mesenchymal Stem Cells Facilitate In Vitro Development of Human Preantral Follicle. Reprod Sci. 2015 Nov;22(11):1367-76. doi: 10.1177/1933719115578922. Epub 2015 Apr 7. PMID 25854744
- [Background] Vural F, Vural B, Doger E, Cakiroglu Y, Cekmen M. Perifollicular blood flow and its relationship with endometrial vascularity, follicular fluid EG-VEGF, IGF-1, and inhibin-a levels and IVF outcomes. J Assist Reprod Genet. 2016 Oct;33(10):1355-1362. doi: 10.1007/s10815-016-0780-7. Epub 2016 Aug 2. PMID 27484063
- [Background] Vahabi S, Yadegari Z, Mohammad-Rahimi H. Correction to: Comparison of the effect of activated or non-activated PRP in various concentrations on osteoblast and fibroblast cell line proliferation. Cell Tissue Bank. 2018 Sep;19(3):455. doi: 10.1007/s10561-017-9677-7. PMID 29270824
- [Background] Pantos K, Nitsos N, Kokkali G, et al. Ovarian rejuvenation and folliculogenesis reactivation in peri-menopausal women after autologous platelet-rich plasma treatment. Abstracts, ESHRE 32nd Annual Meeting; 3-6 Jul 2016; Helsinki, Finland. Hum Reprod 2016 (Suppl. 1):i301.
- [Background] Pines A, Sturdee DW, MacLennan AH. Quality of life and the role of menopausal hormone therapy. Climacteric. 2012 Jun;15(3):213-6. doi: 10.3109/13697137.2012.655923. PMID 22612606
- [Background] Zollner YF, Acquadro C, Schaefer M. Literature review of instruments to assess health-related quality of life during and after menopause. Qual Life Res. 2005 Mar;14(2):309-27. doi: 10.1007/s11136-004-0688-z. PMID 15892422
- [Background] Utian WH, Woods NF. Impact of hormone therapy on quality of life after menopause. Menopause. 2013 Oct;20(10):1098-105. doi: 10.1097/GME.0b013e318298debe. PMID 23799357
- [Background] Hess R, Colvin A, Avis NE, Bromberger JT, Schocken M, Johnston JM, Matthews KA. The impact of hormone therapy on health-related quality of life: longitudinal results from the Study of Women's Health Across the Nation. Menopause. 2008 May-Jun;15(3):422-8. doi: 10.1097/gme.0b013e31814faf2b. PMID 18467950
- [Background] Tella SH, Gallagher JC. Prevention and treatment of postmenopausal osteoporosis. J Steroid Biochem Mol Biol. 2014 Jul;142:155-70. doi: 10.1016/j.jsbmb.2013.09.008. Epub 2013 Oct 29. PMID 24176761
- [Background] Greendale GA, Sowers M, Han W, Huang MH, Finkelstein JS, Crandall CJ, Lee JS, Karlamangla AS. Bone mineral density loss in relation to the final menstrual period in a multiethnic cohort: results from the Study of Women's Health Across the Nation (SWAN). J Bone Miner Res. 2012 Jan;27(1):111-8. doi: 10.1002/jbmr.534. PMID 21976317
- [Background] Samargandy S, Matthews KA, Brooks MM, Barinas-Mitchell E, Magnani JW, Janssen I, Hollenberg SM, El Khoudary SR. Arterial Stiffness Accelerates Within 1 Year of the Final Menstrual Period: The SWAN Heart Study. Arterioscler Thromb Vasc Biol. 2020 Apr;40(4):1001-1008. doi: 10.1161/ATVBAHA.119.313622. Epub 2020 Jan 23. PMID 31969013
- [Background] Greendale GA, Huang M, Cauley JA, Liao D, Harlow S, Finkelstein JS, Hans D, Karlamangla AS. Trabecular Bone Score Declines During the Menopause Transition: The Study of Women's Health Across the Nation (SWAN). J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1872-82. doi: 10.1210/clinem/dgz056. PMID 31613958
- [Background] Randolph JF Jr, Zheng H, Sowers MR, Crandall C, Crawford S, Gold EB, Vuga M. Change in follicle-stimulating hormone and estradiol across the menopausal transition: effect of age at the final menstrual period. J Clin Endocrinol Metab. 2011 Mar;96(3):746-54. doi: 10.1210/jc.2010-1746. Epub 2010 Dec 15. PMID 21159842
- [Background] Burger H. The menopausal transition--endocrinology. J Sex Med. 2008 Oct;5(10):2266-73. doi: 10.1111/j.1743-6109.2008.00921.x. Epub 2008 Jul 1. PMID 18624962
- [Background] Greendale GA, Sternfeld B, Huang M, Han W, Karvonen-Gutierrez C, Ruppert K, Cauley JA, Finkelstein JS, Jiang SF, Karlamangla AS. Changes in body composition and weight during the menopause transition. JCI Insight. 2019 Mar 7;4(5):e124865. doi: 10.1172/jci.insight.124865. eCollection 2019 Mar 7. PMID 30843880
- [Background] Karlamangla AS, Burnett-Bowie SM, Crandall CJ. Bone Health During the Menopause Transition and Beyond. Obstet Gynecol Clin North Am. 2018 Dec;45(4):695-708. doi: 10.1016/j.ogc.2018.07.012. Epub 2018 Oct 25. PMID 30401551
- [Background] Sfakianoudis K, Simopoulou M, Nitsos N, Rapani A, Pappas A, Pantou A, Chronopoulou M, Deligeoroglou E, Koutsilieris M, Pantos K. Autologous Platelet-Rich Plasma Treatment Enables Pregnancy for a Woman in Premature Menopause. J Clin Med. 2018 Dec 20;8(1):1. doi: 10.3390/jcm8010001. PMID 30577435